CLINICAL TRIAL: NCT04599400
Title: Quality and Readability of Online Information on Myofascial Pain Syndrome
Brief Title: Online Information on Myofascial Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Kars State Hospital (Other)
Responsible Party: Principal Investigator, Fatih Bagcier, Principal Investigator, Kars State Hospital
Other Study IDs: Not appropriate
Record Dates: First submitted 2020-10-11; First posted 2020-10-22 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Myofascial Pain Syndrome, Diffuse
Keywords: muscle; pain; online information
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention in our study — There is no intervention in our study

SUMMARY:
The investigators aim in this study is to evaluate myofascial pain syndrome (MPS) related websites in terms of the quality and the readability of the information. Also, to identify the typologies of websites that provide high-quality information about MPS.

DETAILED DESCRIPTION:
Introduction The reliability of information on the internet, which people use as an easy and practical solution about diseases, is very important for public health. The ivestigatior aim in this study to evaluate the quality and readability of websites related to myofascial pain syndrome.

Methods On April 4, 2020, web sites were searched on the Google search engine by using the term "myofascial pain syndrome". The typologies, quality and readability parameters of the sites were analyzed. Websites were divided into eight categories according to typology. In order to evaluate the quality, it is checked whether there is JAMA scoring system and HONcode certificate. Flesch-Kincaid grade and the Simple Measure of Gobbledygook was used to evaluate readability.

ELIGIBILITY:
Inclusion Criteria:

• The URL of the first 200 sites

Exclusion Criteria:

* The sites in languages other than English
* The sites with video and audio recording but without reading text
* The sites with access problems or requesting registration
* Subscription and the sites that do not provide information about myofascial pain syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Not appropriate
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
% of websites | One day
  Websites typologies were commercial (websites that sell or offer a product for profit), government (websites created, administered or regulated by an official government agency), health portal (websites that provide information about health issues), news (news and information created to provide newspaper or magazine websites), non-profit (charitable/supportive/educational websites that were not established for the purpose of profit-making), professional (websites created by organizations or individuals with professional medical qualifications), scientific journal (accessible scientific articles or academic publications). Websites that do not fit any typology were categorized under the heading of others.
Readability Scores | One day
  The investigators used an online tool to assess the Flesch-Kincaid Grade. The "FKG Level Formula" presents a score as a US grade level, thereby making it easier for teachers, parents, librarians, and others to judge the readability level of various books and texts. The FKG evaluates the average sentence length and average syllables per word in the calculation of readability score The investigators used an online tool to assess the Flesch-Kincaid Grade (FKG) scores of websites (https://www.webfx.com/tools/read-able/).
  The "FKG Level Formula" presents a score as a US grade level, thereby making it easier for teachers, parents, librarians, and others to judge the readability level of various books and texts. The FKG evaluates the average sentence length and average syllables per word in the calculation of readability score
Readability Scores | One day
  The investigators used an online tool to assess the Simple Measure of Gobbledygook (SMOG) scores of websites (https://www.webfx.com/tools/read-able/).
  The SMOG grade is a measure of readability that estimates the years of education needed to understand a piece of writing. In addition to parameters in the FKG scoring system, the SMOG grade evaluates the number of polysyllabic words in 30 sentences. The SMOG is widely used, particularly for checking health-related texts.
  The SMOG readability formula consists of a readability equation based on average sentence length and 3 or more syllable word ratio variables
Quality Scores | One day
  It consists of four parts;
  1. Authorship; In this section, the authors, contributors and their identity information and the institutions they are affiliated with must be specified.
  2. Bibliography; All sources and references must be listed; copyright must be specified.
  3. Patent right; The "ownership" of the website must be clearly and fully disclosed, with sponsorship, advertising, insurance, business support and potential conflicts of interest.
  4. Actuality; The date when the content was published and updated must be specified.
  Evaluations were made by giving 1 point to each item meeting these criteria. The lowest score that can be obtained in the JAMA criteria is "0" and the highest score is 4. A website with ≥3 points is considered as high quality, whereas ≤2 is considered as low quality. Two independent investigators (FB and OVY) evaluated JAMA scores.
Reliability sertification | One day
  The Health on the Net Foundation (HON), established to promote the online delivery of useful and reliable health information and to ensure its convenient and efficient use, has prepared HONcode to help standardize the reliability of health information available on the web.
  HONcode criteria; authors' competencies should be stated, patient-physician should complete the relationship, the privacy policy should be explained, the source and date of the content should be explained, the content should be compared, the contact information should be explained, the financing of the site should be explained, and the advertisement policy should be explained. HON issues the HONcode compliance certificate to the evaluated websites. If HONcode is available on the website, that website can be considered a high quality website.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Bagcier, Principal Investigator — Biruni University Faculty of Medicine
Locations (1):
- Biruni University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No